CLINICAL TRIAL: NCT05192837
Title: Preoperative Smoking Cessation Program in Patients Undergoing Intermediate to High-risk Surgery: a Randomized, Single-blinded, Controlled Trial
Brief Title: Preoperative Smoking Cessation in Patients Undergoing Surgery
Acronym: PORTICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Christian Fankhauser, Principal Investigator, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-8131
Record Dates: First submitted 2022-01-01; First posted 2022-01-14 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation; Smoking Reduction; Surgery--Complications; Surgery; Cancer; Postoperative Complications; Perioperative Complication; Smoking; Abdominal Cancer; Thoracic Cancer; Urologic Cancer; Gynecologic Cancer; Head and Neck Cancer
Keywords: preoperative smoking cessation; intensive smoking cessation; intermediate-risk surgery; high-risk surgery; nicotine replacement therapy; varenicline; bupropion; clavien dindo classification; comprehensive complication index; epic; electronic health record
MeSH Terms: conditions — Smoking Cessation; Smoking Reduction; Neoplasms; Postoperative Complications; Smoking; Urologic Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 1:1 ratio to either the intervention or control group using service of the University of Graz (www.randomizer.at). Before randomisation patients will be pre-stratified for age (≤60, >60 years) and procedure (intermediate versus high-risk procedures). Both factors have been identified in a previous retrospective cohort study at our institution as risk factors for complications. For that reason, minimization, as an efficient way to control for confounding in small to moderately sized trials, will be used. Also, minimization automatically ensures concealment of random allocation since there is no pre-existing randomization list.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Throughout the study patient data is collected in the electronic health record (LUKiS) in an uncoded manner. Allocation will be blinded. At the end of the study the LUKiS reporting team will generate a report, which will include all study data in a de-identified form. The analysis of the report with the pseudonymized data will be performed by the project statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The study intervention consists of a smoking cessation counselling meeting by a Tabacco Treatment Specialist (TSS) 4 weeks before surgery. The goal of this first intervention meeting is to implement an individual treatment plan for preoperative smoking cessation.
  Interventions: Behavioral: Intensive preoperative smoking cessation counselling
- Control group (No Intervention): Patients randomised to the control arm will get advice only. Their preoperative course will be as if they were not participating in this study, meaning they will receive inconsistent perioperative smoking cessation advice from nurses, surgeons, or anaesthesiologists but no further study-specific smoking cessation intervention. Importantly, participants in the control group will not be discouraged from using perioperative smoking cessation aids and can still obtain help on one's own initiative.

INTERVENTIONS:
Behavioral: Intensive preoperative smoking cessation counselling — The study intervention consists of an interview by a Tabacco Treatment Specialist (TSS) 4 weeks before surgery with individual counselling and offered nicotine substitution. The intervention meeting is based on the Chronic Care Model (CCM) to improve quality of ambulatory care.
  In brief, the intervention includes:
  * Informative content about advantages of smoking cessation
  * Scheduling service for a motivational interview by a TSS in office to implement a treatment plan
  * For participants willing to quit smoking a preoperative quit day will be scheduled after the first intervention meeting 2-3 weeks before surgery
  * Patients will be encouraged by a TSS to use nicotine replacement. Bupropion or Vareniclin will be provided on an individual basis
  * TSS will schedule repeated follow-up meetings to support smoking abstinence or nicotine reduction before and after surgery for all patients
  Arms: Intervention group

SUMMARY:
Background: At present, effectively implementing smoking cessation programs in the health care system constitutes a major challenge. A unique opportunity to initiate smoking cessation focuses on smokers scheduled for surgery. These patients are not only highly motivated to quit smoking but also likely to benefit from a reduction in postoperative complications which may translate into a decrease of costs. Nevertheless, surgical patients are not routinely informed about the benefits of preoperative smoking cessation. Potential reasons for this missed opportunity may be lack of time and training of surgeons and anesthesiologists. The investigators therefore aim to analyse the impact of a preoperative high-intensity smoking cessation intervention on surgical complications up to a 90-day postoperative period in patients of various surgical disciplines. The hypothesis is that preoperative smoking cessation program improves outcomes in smokers undergoing intermediate to high-risk surgery. The primary objective is to compare complications between patients with an institutional multifaceted smoking cessation intervention starting four weeks before surgery compared to patients in the advice only group (control group) within a 90-day postoperative period. The primary endpoint is the Comprehensive Complication Index (CCI®) within 90 days of surgery. Secondary outcomes include length of hospital stay, cost of hospital stay, smoking abstinence, reduction in nicotine consumption.

Methods: The present study is a single center, randomized trial with two parallel groups of smokers scheduled for surgery comparing surgery alone and surgery with preoperative smoking cessation. The investigators plan to randomize 251 patients. The primary endpoint is the Comprehensive Complication Index up to a 90-day postoperative period. The secondary endpoints include comparison of smoking abstinence, quality of life, mental health, length of stay, costs of care and difference in hospital reimbursement between the two groups.

Discussion: The hypothesis is that preoperative smoking cessation program improves outcomes in smokers undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient listed for intermediate or high-risk surgery at the Kantonsspital of Lucerne
* Patient undergoing surgery in one of the following departments: Abdominal surgery, thoracic surgery, cardiac surgery, urology, gynaecology, vascular surgery or head and neck surgery
* Date of surgery >2 weeks after date of listing for surgery or discussion by tumor board
* Current smokers, defined as daily smoking of at least one cigarette, cigar or pipe
* Age over 18 years
* Able to give signed written informed consent

Exclusion Criteria:

* Plastic surgery
* Consumption of illegal drugs
* Alcohol dependency defined as preexisting alcohol related disorders (eg. alcoholic psychosis, Alcohol abuse, Alcohol polyneuropathy, degeneration of nervous system due to alcohol, Alcoholic myopathy, Alcoholic liver disease)
* Inability to follow the procedures of the study, e.g., due to language problems, psychological disorders, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index (CCI) | within a 90 days postoperative time period
  The primary endpoint is the Comprehensive Complication Index (CCI) within 90 days of surgery. The CCI is calculated as the sum of all Clavien-Dindo complications that are weighted for their severity (multiplication of the median preference values from patients and physicians). The final formula yields a continuous scale that ranks the cumulative burden from any combination of complications from 0 to 100 with higher values indicating a higher cumulative burden in a single patient. As a composite complication score, the CCI has the advantage of reflecting the overall burden of the postoperative course that affects the health of patients and their quality of life. In addition, the CCI is a powerful endpoint in trials, as it allows sample size up to nine times lower compared with traditional morbidity endpoints.

SECONDARY OUTCOMES:
Length of hospital stay | perioperative
  Days of hospital stay for planned surgery
Costs of hospital stay | perioperative
  Costs of hospital stay for planned surgery
Readmission rate | within a 90 days postoperative time period
  Readmission rates for in-patient hospital stay after surgery
Smoking abstinence | within a one year postoperative time period
  Number of patients who successfully quit smoking
Smoking reduction | within a one year postoperative time period
  Decrease or increase of daily nicotine consumption
Mental health | one week preoperative
  The outcome is measured using the Hospital anxiety and depression scale (HADS) before surgery. The score ranges from 0 to 42 with higher values indicating a higher probability of a mood disorder.
IMC/ICU admission | perioperative
  unplanned postoperative intermediate care or intensive care unit admission
Transtheoretical Model | preoperative
  Stage of the Transtheoretical Model of behaviour change
Quality of life Short Form Survey | within a one year postoperative time period
  The outcome is measured using the 36-Item Short Form Survey (SF-36). The score ranges from 0 to 100 with higher values indicating a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Fankhauser, PD Dr. med., Principal Investigator — Klinik für Urologie, Luzerner Kantonsspital
Locations (1):
- LUKS, Lucerne, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fankhauser CD, Affentranger A, Cortonesi B, Jeker U, Gass M, Minervini F, Jung G, Christmann C, Brambs C, Puhan MA, Held U. Preoperative smoking cessation program in patients undergoing intermediate to high-risk surgery: a randomized, single-blinded, controlled, superiority trial. Trials. 2022 Aug 29;23(1):717. doi: 10.1186/s13063-022-06628-8. PMID 36038883